CLINICAL TRIAL: NCT07240571
Title: Family-Focused Adolescent & Lifelong Health Promotion: Prevention of Adolescent Mental Health Problems in Eastern Europe
Brief Title: Randomized Controlled Trial of a Family-focused Intervention for Caregivers and Young Adolescents (Phase 3 of FLOURISH)
Acronym: FLOURISH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Klagenfurt (Other)
Collaborators: Health for Youth Association, Moldova (Other); Institute for Marriage, Family and Systemic Practice - ALTERNATIVA (Other); Cardiff University (Other); Medical University of Vienna (Other); Bielefeld University (Other); University Jaume I Castellon (Unknown); Association of Systemic Therapists Education Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20230135
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Adolescent - Emotional Problem; Parent Child Relationship; Family Functioning; Well-Being, Psychological
Keywords: Multiphase Optimization Strategy (MOST); Family-based intervention; Adolescents; Mental health; Randomized trial
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimized Parenting for Lifelong Health (PLH) for Parents and Teens (Experimental): Families assigned to this arm will receive the optimized Parenting for Lifelong Health (PLH) for Parents and Teens program. The intervention is delivered in groups of approximately 10 adolescent-caregiver pairs over a 7-week period. It includes one pre-program visit and six weekly group sessions (about two hours each), with a mix of joint and separate sessions for caregivers and adolescents. Sessions are facilitated by trained professionals under ongoing supervision to ensure fidelity. The program focuses on strengthening family relationships, improving communication, managing emotions, problem-solving, and promoting positive parenting.
  Interventions: Behavioral: Optimized Parenting for Lifelong Health (PLH) for Parents and Teens
- Waitlist Control (No Intervention): Families assigned to this arm will not receive the intervention during the initial study period. They will complete all study assessments at baseline, post-intervention, and 6-month follow-up. After completion of the 6-month follow-up assessment, families in the waitlist control arm will be offered the optimized Parenting for Lifelong Health (PLH) for Parents and Teens program under the same delivery format as the intervention group.

INTERVENTIONS:
Behavioral: Optimized Parenting for Lifelong Health (PLH) for Parents and Teens — The optimized Parenting for Lifelong Health (PLH) for Parents and Teens program is a group-based parenting and adolescent skills training intervention. It will be delivered to adolescent-caregiver pairs (ages 10-14 and their primary caregivers) in groups of about 10 families. The program lasts 7 weeks and includes one pre-program visit and six weekly group sessions of approximately two hours each. Sessions include both joint and separate modules for caregivers and adolescents, focusing on building positive relationships, managing emotions, establishing routines, problem solving, and strengthening family communication. The program is facilitated by trained professionals who receive two days of training and ongoing weekly supervision.
  Arms: Optimized Parenting for Lifelong Health (PLH) for Parents and Teens

SUMMARY:
The aim of this study is to conduct a multi-country randomized waitlist controlled trial to evaluate the effectiveness, cost-effectiveness, and scalability of the optimized Parenting for Lifelong Health (PLH) for Parents and Teens program in Moldova and North Macedonia. In Phase 2 of the FLOURISH project, a factorial trial tested multiple intervention components and identified the optimized intervention package. In Phase 3, this trial will assess the implementation, outcomes, and economic impact of the optimized PLH program delivered to adolescents aged 10-14 and their caregivers. ALTERNATIVA will deliver the program in North Macedonia and the Health for Youth Association in the Republic of Moldova.

DETAILED DESCRIPTION:
Adolescent mental health is a significant global concern, especially in low- and middle-income countries (LMICs) like North Macedonia and Moldova. Adolescents in LMICs face numerous challenges, including socio-economic stressors, adverse childhood experiences, and limited access to mental health services. Parenting interventions are one approach to reduce risk for poor adolescent mental health outcomes and family maltreatment. Systematic evaluation of parenting programs is essential for enhancing scalability and sustainability in low-resource settings.

Building on prior research, the Family-Focused Adolescent & Lifelong Health Promotion (FLOURISH) project aims to adapt, optimize, and evaluate a parenting intervention for adolescents aged 10-14 and their caregivers in North Macedonia and Moldova. The project focuses on improving adolescent mental health and well-being in both teens and caregivers, and it is implemented according to the Multiphase Optimization Strategy (MOST) framework.

Phase 1 of the project assessed the feasibility and cultural adaptation of the PLH for Parents and Teens program. In Phase 2, a multi-country factorial trial tested different combinations of three additional components (adolescent mental health tools from UNICEF's Helping Adolescents Thrive comics, adolescent peer support, and engagement boosters) and identified the optimized intervention package.

This protocol describes the evaluation (Phase 3) of the optimized FLOURISH intervention package. The randomized waitlist controlled trial will recruit adolescent-caregiver pairs (320 to 340 families per country, 640 to 660 total) to test the effectiveness, cost-effectiveness, and scalability of the optimized PLH program. Families assigned to the intervention group will receive the program over seven weeks (one pre-program visit and six weekly group sessions), while families in the waitlist control group will receive the intervention after the six-month follow-up assessment. The results of this study will inform the potential for scaling up the optimized intervention at the national level in both countries and contribute robust evidence on adolescent mental health promotion in LMICs.

ELIGIBILITY:
Inclusion Criteria:

* For Caregivers:

Must be 18 years or older at baseline assessment

Must be the primary caregiver of an adolescent aged 10-14 who has resided in the same household for at least four nights a week in the past month

Must be able to speak at least one of the local languages in which the program will be offered (e.g., Macedonian, Romanian, Russian, Ukrainian or Albanian)

Must agree to participate in the program and provide informed consent for both themselves and their adolescent

For Adolescents:

Must be aged 10-14 at the baseline assessment

Must provide assent to participate in the study

Must have caregiver consent to participate.

Exclusion Criteria:

* No formal exclusion criteria have been established for the FLOURISH project. However, during the study introduction, the research team will guide participants through a consent form that asks whether they are currently experiencing acute distress or a mental or physical health condition that could interfere with participation. The decision to participate will be made by the individual. If a potential participant indicates they are unable to take part due to acute health issues, the research team will provide appropriate referrals to other services.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1280 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in levels of emotional and behavioral problems in adolescents (caregiver report): Pediatric Symptom Checklist (PSC-17), internalizing subscale | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The PSC-17 (caregiver-report) includes 17 items, with responses from 0 (never) to 2 (often) and assesses adolescents' psychosocial functioning. The internalizing subscale includes 5 items. Higher scores indicate more emotional problems.
Change in levels of family functioning in caregivers: Family Assessment Device (FAD), subscale general functioning | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The general functioning subscale is one of the dimensions of the FAD and will be completed by caregivers. It consists of 12 items. Scoring is on a 4-point scale (from 1 = strongly agree to 4 = strongly disagree). Higher scores indicate poorer family functioning.
Change in frequency of parenting practices in caregivers (caregiver-report): Alabama Parenting Questionnaire (APQ), subscales involved and positive parenting | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  Parenting practices will be assessed with the caregiver-report version of the APQ. The APQ is a self-report measure of parenting behaviors designed to assess practices most related to children's behavioral adjustment. Items are rated on a 5-point scale from 1 (never) to 5 (always). Higher scores on the involved and positive parenting subscales indicate more positive parenting practices. It is completed by caregivers.
Change in caregiver health-related quality of life: EQ-5D-5L | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The EQ-5D-5L is a standardized instrument developed to measure health-related quality of life. It consists of five dimensions, each rated on a 5-point scale: no problems, slight problems, moderate problems, severe problems, and extreme problems. Additionally, it includes a visual analogue scale (VAS) ranging from 0 (worst imaginable health) to 100 (best imaginable health). Higher dimension scores indicate more health problems; higher VAS scores indicate better self-rated health. It is completed by caregivers.
Change in adolescent health-related quality of life: EQ-5D-Y-3L | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The EQ-5D-Y-3L is a standardized instrument designed to measure health-related quality of life in children and adolescents. It consists of five dimensions, each rated on a 3-point scale: no problems, some problems, severe problems. It also includes a visual analogue scale (VAS) from 0 (worst imaginable health) to 100 (best imaginable health). Higher dimension scores indicate more health problems; higher VAS scores indicate better self-rated health. It is completed by adolescents.

SECONDARY OUTCOMES:
Change in levels of family communication in adolescents: Child-Parent Communication Apprehension scale (CPA-YA), total score | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The CPA-YA measures parent-child communication apprehension and is completed by adolescents. Each item is scored on a 5-point Likert scale (0 = strongly agree to 4 = strongly disagree). Four items are reverse-coded so that all responses are oriented in the same direction. Higher scores indicate less communication apprehension (i.e., more ease and confidence in communicating with parents).
Change in levels of loneliness in adolescents: UCLA-8 Loneliness scale, total score | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The UCLA-8 is an 8-item scale designed for adolescents. Items are rated on a 4-point scale (1 = never to 4 = often). Higher scores indicate greater loneliness.
Change in frequency of parenting practices (adolescent-report): Alabama Parenting Questionnaire (APQ), subscales involved and positive parenting | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The APQ adolescent-report version measures perceptions of parenting behaviors. Items are rated on a 5-point scale from 1 (never) to 5 (always). Higher scores on involved and positive parenting subscales indicate better parenting practices.
Change in levels of emotional and behavioral problems in adolescents (adolescent-report): Pediatric Symptom Checklist (PSC-17), internalizing, externalizing and attention subscales, total score | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The PSC-17 (adolescent-report) includes 17 items with a response range from 0 (never) to 2 (often), assessing overall psychosocial problems. Higher scores indicate more emotional and behavioral problems.
Change in levels of well-being in adolescents: World Health Organization-Five Well-Being Index (WHO-5), total score | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The WHO-5 includes 5 items rated from 0 (none of the time) to 5 (all of the time), assessing subjective well-being over the past 14 days. Scores range from 0 (lowest well-being) to 25 (highest well-being). Higher scores indicate greater well-being. It is completed by adolescents.
Change in levels of emotional problems in adolescents: Revised Child Anxiety and Depression Scale (RCADS), depression and anxiety subscales, total score | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The RCADS (adolescent self-report) consists of 25 items, each rated on a 4-point Likert scale (0 = never, 1 = sometimes, 2 = often, 3 = always). Item responses are summed to create separate scores for anxiety, depression, and a total score. Higher scores indicate greater anxiety, depressive symptoms, and overall emotional problems.
Change in adolescent socio-emotional skills: Social Emotional Abilities and Learning (SEAL) Tool, subscales emotional regulation, problem-solving, interpersonal skills | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The SEAL emotional regulation, problem-solving, interpersonal skills subscales include 7 items with responses "yes," "no," or "maybe." Higher scores indicate better socio-emotional skills. The questionnaire is completed by adolescents.
Change in levels of bullying involvement in adolescents: Health Behaviour in School-aged Children (HBSC), peer violence subscale | Pre-assessment and 6-month follow-up
  The HBSC bullying module captures both traditional and cyber forms of bullying, including victimization and perpetration, over the past couple of months. It consists of 4 items covering bullying others, being bullied, cyberbullying perpetration, and cyberbullying victimization. Each item is scored on a 5-point scale: 0 = not in the past couple of months, 1 = once or twice, 2 = 2-3 times a month, 3 = about once a week, 4 = several times a week. Higher scores indicate greater involvement in bullying or cyberbullying. It is completed by adolescents.
Change in levels of parent-child communication in adolescents: Parent-Child Communication scale | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The Parent-Child Communication scale (adolescent-report) consists of 7 items assessing the adolescent's ability to communicate feelings, problems, and beliefs with their caregiver. Items are rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate better communication between the adolescent and caregiver.
Change in levels of social support in adolescents: Medical Outcome Study Social Support Survey (MOS-SSS), emotional and affectionate subscales | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The MOS-SSS includes 18 items with a response range from 1 (none of the time) to 5 (all of the time). The emotional and affectionate subscales together comprise 11 items. Higher scores indicate greater perceived social support. It is completed by adolescents.
Change in frequency of parenting practices in caregivers: Alabama Parenting Questionnaire (APQ), subscale corporal punishment | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The APQ caregiver-report version measures frequency of disciplinary practices. Items are rated on a 5-point scale from 1 (never) to 5 (always). Higher scores on the corporal punishment subscale indicate greater use of punitive parenting practices. It is completed by caregivers.
Change in frequency of emotionally maltreating behaviors in caregivers: International Child Abuse Screening Tool (ICAST), emotional maltreatment subscale | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  This subscale consists of 5 items assessing psychologically aggressive behaviors toward the child in the past 4 weeks, including verbal aggression, emotional shaming, withdrawal, and threats of abandonment. Each item is scored on a 9-point frequency scale (0 = never to 8 = 8 or more times). Higher scores indicate greater frequency of emotional maltreatment.
Change in levels of well-being in caregivers: World Health Organization-Five Well-Being Index (WHO-5), total score | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The WHO-5 includes 5 items rated from 0 (none of the time) to 5 (all of the time), assessing subjective well-being over the past 14 days. Scores range from 0 (lowest well-being) to 25 (highest well-being). Higher scores indicate greater well-being. It is completed by caregivers.
Change in levels of psychological distress in caregivers: Patient Health Questionnaire-9 (PHQ-9), total score | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The PHQ-9 is a 9-item self-report tool for depressive symptom severity. Items are scored from 0 (not at all) to 3 (nearly every day). Higher scores indicate more depressive symptoms. It is completed by caregivers.
Change in levels of parental stress in caregivers: Parental Stress Scale (PSS), total score | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The PSS is an 18-item self-report questionnaire rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Higher scores indicate greater parental stress. It is completed by caregivers.
Change in levels of loneliness in caregivers: Revised UCLA Loneliness Scale (RULS-6), total score | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The RULS-6 consists of 6 items rated on a Likert scale (from 1 = never to 4 = always). Item responses are summed to create a total score ranging from 6 to 24, with higher scores indicating greater loneliness. It is completed by caregivers.
Change in levels of social support in caregivers: Medical Outcome Study Social Support Survey (MOS-SSS), emotional and affectionate subscales | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The MOS-SSS emotional and affectionate subscales comprise 11 items. Scores range 1 (none of the time) to 5 (all of the time). Higher scores indicate more perceived social support. It is completed by caregivers.
Change in levels of family functioning in caregivers: Family Assessment Device (FAD), problem solving subscale | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The problem solving subscale (6 items) assesses ability to resolve problems. Responses range from 1 (strongly agree) to 4 (strongly disagree). Higher scores indicate poorer functioning. It is completed by caregivers.
Change in caregiver capabilities: Oxford CAPabilities questionnaire - Mental Health (OxCAP-MH), total score | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The OxCAP-MH includes 16 items across domains such as social participation, emotional stability, and access to resources. Items are scored on a 5-point Likert scale. It is completed by caregivers.
Change in caregiver resource use: PECUNIA Resource Use Measurement (PECUNIA RUM) | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The PECUNIA RUM assesses caregivers' use of residential care, non-residential health and social care, informal help, and work-related resources.
Change in caregiver-reported resource use in adolescents (caregiver-report): PECUNIA Resource Use Measurement (PECUNIA RUM) | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The PECUNIA RUM proxy for adolescents records service use reported by caregivers, covering residential care, non-residential health and social care, and education.
Change in levels of parent-child communication in caregivers: Parent-Child Communication Scale | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The Parent-Child Communication Scale (caregiver-report) includes 7 items assessing caregiver perceptions of openness, emotional expressiveness, problem discussion, and perspective-taking in communication with their child. Items are rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Total scores range from 7 to 35. Higher scores indicate more open, emotionally supportive, and bidirectional communication.
Change in levels of emotional and behavioral problems in adolescents (caregiver-report): Pediatric Symptom Checklist (PSC-17), externalizing and attention subscales, total score | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The PSC-17 (caregiver-report) includes 17 items with a response range from 0 (never) to 2 (often), assessing overall psychosocial problems. The externalizing and attention subscales include 12 items. Higher scores indicate more emotional and behavioral problems.

OTHER OUTCOMES:
Adolescent healthy weight: Body Mass Index (BMI), adolescent-report | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  BMI will be calculated from adolescent-reported mass (kg) and height (m).
Adolescent healthy weight: Body Mass Index (BMI), caregiver-report | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  BMI will also be calculated from caregiver-reported adolescent mass (kg) and height (m).
Post-traumatic stress in caregivers: PTSD Checklist for DSM-5 (PCL-5), short form, total score | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The short form of the PCL-5 includes 4 items assessing PTSD symptom severity. Each item is scored from 0 (not at all) to 4 (extremely), with higher scores indicating greater PTSD symptoms. It is completed by caregivers.
Well-being among intervention staff: World Health Organization-Five Well-Being Index (WHO-5), total score | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The WHO-5 is a brief measure of emotional well-being over the past 14 days. It includes 5 items scored from 0 (none of the time) to 5 (all of the time). Total scores range from 0 (absence of well-being) to 25 (maximum well-being). Higher scores indicate greater well-being. It is completed by intervention staff.
Fidelity of intervention delivery: PLH-Facilitator Assessment Tool (PLH-FAT) | During intervention implementation (6-8 weeks)
  The PLH-FAT evaluates fidelity of intervention delivery based on facilitator performance. It yields percentage scores on completion of intervention activities and demonstration of intervention skills. Higher percentages indicate greater fidelity.
Intervention costs | During intervention implementation (6-8 weeks)
  Intervention costs will include personnel time for training and delivery, organizational costs, materials, transportation, and consumables.
Caregiver-defined problems on the adolescent: Top Problems Assessment (TPA) | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The TPA allows caregivers to identify their adolescent's three most pressing emotional or behavioral problems and rate each on a scale from 0 (not a problem) to 4 (a very big problem). Higher scores indicate greater severity of caregiver-identified problems.
Adolescent-defined problems: Top Problems Assessment (TPA) | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The TPA allows adolescents to identify their three most important problems and rate each on a scale from 0 (not a problem) to 4 (a very big problem). Higher scores indicate greater severity of self-identified problems.
Attendance rate | During intervention implementation (6-8 weeks)
  Attendance will be assessed for: individual attendance, defined as the percentage of PLH sessions out of six attended separately by adolescents and caregivers; family attendance, defined as the percentage of PLH sessions out of six attended jointly by both adolescent and caregiver; and catch-up attendance, defined as the percentage of scheduled catch-up sessions attended out of six. Higher percentages indicate greater attendance.
Enrollment rate | During intervention implementation (6-8 weeks)
  Enrollment will be assessed as: individual enrollment, measured as the percentage of adolescents and caregivers who attended at least one PLH session; family enrollment, measured as the percentage of families in which both the adolescent and caregiver attended at least one PLH session. Higher percentages indicate greater enrollment.
Parenting among intervention staff: Alabama Parenting Questionnaire (APQ), involved and positive parenting subscales | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The APQ is a self-report instrument of parenting practices. The involved and positive parenting subscales each assess positive caregiver behaviors such as engagement, attention, and supportive interactions. Items are rated on a 5-point scale ranging from 1 (never) to 5 (always). Higher scores indicate more positive and involved parenting practices.
Post-traumatic stress in adolescents: Children's Revised Impact of Event Scale (CRIES), total score, intrusion and avoidance subscales | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The CRIES includes 8 items, scored on a 4-point scale (0 = not at all, 1 = rarely, 3 = sometimes, 5 = often). It provides a total score and two subscales: intrusion and avoidance. Higher scores indicate greater trauma-related distress. It is completed by adolescents.
Changes in levels of food insecurity in caregivers: Food Insecurity Experience Scale (FIES) | Pre-assessment, 8-12 weeks after pre-assessment, and 6-month follow-up
  The FIES consists of 8 items assessing household experiences of food insecurity in the past 12 months, from worry about food availability to skipping meals or going a whole day without eating due to lack of money or resources. Items are scored yes (1) or no (0). Higher scores indicate more severe food insecurity. It is completed by caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Foran, Prof, Principal Investigator — University of Klagenfurt; Yulia Shenderovich, Dr, Principal Investigator — Cardiff University; Marija Raleva, Principal Investigator — Institute for Marriage, Family and Systemic Practice - ALTERNATIVA; Galina Dr Lesco, Principal Investigator — Health for Youth Association, Moldova; Graham Moore, Prof, Principal Investigator — Cardiff University; Rhiannon Evans, Prof, Principal Investigator — Cardiff University; Judit Simon, Prof, Principal Investigator — Medical University of Vienna; Nina Heinrichs, Prof, Principal Investigator — Bielefeld University; Nevena Calovska, Prof, Principal Investigator — Association of Systemic Therapists Education Centre; Bojan Shimbov, Prof, Principal Investigator — University Jaume
Locations (2):
- Health For Youth Association, Chisinau, Moldova
- Institute for Marriage, Family and Systemic Practice - ALTERNATIVA, Skopje, North Macedonia

IPD SHARING:
Plan to Share IPD: Yes
The project has a detailed data management plan (DMP) that defines data sharing procedures. The DMP was provided as a deliverable to the European Commission and is updated throughout the study funding period.
Supporting Information: Study Protocol
Time Frame: After completion of the study and publication of the main results
Access Criteria: Prof. Heather Foran is responsible for data management of the FLOURISH project. For information related to data sharing, please contact her at heather.foran@aau.at
URL: https://www.flourish-study.org